CLINICAL TRIAL: NCT02012452
Title: Tobacco Treatment as Augmentation to Cognitive Processing Therapy for PTSD
Brief Title: Tobacco Treatment as Augmentation for Cognitive Processing Therapy for PTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moving outside VA- grant not transferable
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NURA-018-13S; 1IK2CX000918-01A1 (NIH)
Record Dates: First submitted 2013-09-26; First posted 2013-12-16 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Posttraumatic Stress Disorder; Tobacco Dependence
Keywords: posttraumatic stress disorder; tobacco dependence; cognitive behavioral therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tobacco treatment (Experimental): participants will be provided contingency management and cognitive behavioral therapy to help them quit tobacco prior to PTSD treatment
  Interventions: Behavioral: Tobacco treatment
- health education treatment (Sham Comparator): Participants will be provided education on a variety of health topics and will set health goals around each topic
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Tobacco treatment — participants will be provided contingency management and cognitive behavioral therapy to help them quit tobacco prior to PTSD treatment
  Arms: tobacco treatment
Behavioral: Health Education — Participants will be provided education on a variety of health topics and will set health goals around each topic
  Arms: health education treatment

SUMMARY:
The purpose of this study is to examine whether tobacco affects recovery from PTSD. There are 3 goals of the study; (1) to test if quitting tobacco prior to PTSD treatment affects treatment success, (2) to test how PTSD symptoms change in those who have quit tobacco compared to those who continue to use and (3) to explore how tobacco use and tobacco withdrawal symptoms change during PTSD treatment.

DETAILED DESCRIPTION:
The proposed research aims to examine the effect of tobacco on PTSD symptoms and PTSD recovery as well as the effect of PTSD recovery on tobacco use. This study has 3 aims: (1) to evaluate whether tobacco use interferes with recovery from PTSD during empirically based, trauma focused PTSD treatment. (2) To gather preliminary data about whether tobacco use alleviates PTSD symptoms among continued tobacco users vs. recent quitters. (3) To explore the impact of recovery from PTSD treatment on tobacco use quantity and frequency, tobacco withdrawal symptoms, and craving for tobacco. To test these aims, the investigators propose a randomized two group design where 75 participants are assigned to receive either tobacco treatment (Contingency Management plus Cognitive Behavioral Therapy) or control treatment (Health Education) before completing Cognitive Processing Therapy (CPT) for PTSD. Study outcome variables will be PTSD symptom severity following CPT, PTSD symptom severity during tobacco cessation treatment, and tobacco use and tobacco withdrawal during CPT.

ELIGIBILITY:
Inclusion Criteria:

* current tobacco use (a urine cotinine level 200ng/ml),
* motivation to quit (measured by the 7 on the Biener Contemplation ladder)
* and a current diagnosis of PTSD [as diagnosed by the Clinician Administered PTSD Scale for DSM-5]

Exclusion Criteria:

* Exclusion criteria will include current participation in another research study, history of bipolar I disorder,
* schizophreniform disorders except for psychosis NOS due to presence of trauma-related sensory hallucinations,
* cognitive impairment (<25 of the Mini Mental State Exam),
* current suicidality/homicidality requiring clinical intervention or a suicide attempt in the past year,
* inability to provide reliable study data (e.g., provide an adulterated urine sample,
* provide misinformation to study staff including stating differing information to two or more staff members,
* attempt to misrepresent self in order to avoid being excluded from the study,
* inability to answer study questions which are used to determine eligibility),
* current non-tobacco substance use disorder (abuse or dependence or a positive drug screen; participants who have been abstinent for greater than 3 months will be allowed to participate),
* participation within the past 6 months in trauma-focused therapy (e.g., Prolonged Exposure, Cognitive Processing Therapy),
* current use of tobacco cessation pharmacotherapy (i.e., nicotine replacement therapy or varenicline),
* current use of benzodiazepines
* serious or uncontrolled medical condition precluding unaided tobacco cessation attempts,
* pregnancy,
* a recent change in psychiatric medications (change occurred <2 months prior to entering the study),
* current participation in another research study.
* In addition, participants must agree to keep psychiatric medication doses stable for the duration of the study (except for dose adjustments for changes in medication blood levels due to tobacco cessation), unless there is a concern for participant safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Japuntich, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 participants came in for an in-person screening visit. Of those, 9 met inclusion criteria.
Period: Overall Study
Arm/Group | Tobacco Treatment | Health Education Treatment
Started | 7 | 2
Completed | 1 | 1
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobacco Treatment | Health Education Treatment | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.35 (7.24) | 57.05 (9.66) | 57.12 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 2 | 9
Clinical Administered PTSD scale [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-80. Higher scores indicate greater PTSD severity.
  units on a scale | 40.86 (14.51) | 50.0 (8.49) | 42.89 (13.53)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale
Description: posttraumatic stress disorder clinician rated symptom ratings; scores range from 0-80 (with higher scores indicating greater PTSD severity)
Time Frame: end of 6 week PTSD treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tobacco Treatment | Health Education Treatment
Number analyzed (Participants) | 2 | 1
units on a scale | 18.67 (8.33) | 12 (0)

2. Secondary Outcome: Percent Abstinent From Tobacco Use
Description: biochemically confirmed abstinence from tobacco using self-report, cotinine, and CO breath samples
Time Frame: end of treatment
Population: If participants did not come the follow-up visit they were assumed to be smokers. If they attended a later follow-up visit, tobacco use was retroactively assessed.
Measure: Number; unit: percent abstinent
Arm/Group | Tobacco Treatment | Health Education Treatment
Number analyzed (Participants) | 7 | 2
percent abstinent | 14.3 | 0

ADVERSE EVENTS:
Time Frame: 25 months
Arm/Group | Tobacco Treatment | Health Education Treatment
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/2
Other Adverse Events (participants affected / at risk) | 1/7 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tobacco Treatment (N=7) | Health Education Treatment (N=2)
hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) — Participant went to the ER for chest pain but it was diagnosed as reflux
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tobacco Treatment (N=7) | Health Education Treatment (N=2)
psychosis (Psychiatric disorders) | 1 (1) | 0 (0) — participant was reporting some delusions (e.g., that the therapist could tell the government to change the laws because the VA is part of the government) the participant later tested positive for cocaine at this visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes